CLINICAL TRIAL: NCT02760173
Title: Verticality Perception - Effects of Prolonged Roll-tilt in Healthy Human Subjects
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This protocol was re-written and resubmitted under a different trial number again (NCT02980419)
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: vert_perc_posttilt
Record Dates: First submitted 2016-04-26; First posted 2016-05-03 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Vestibular; Perception
Keywords: verticality perception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single intervention arm (Experimental): This is the only arm in this study, measuring verticality perception after prolonged roll-tilt over 5min.
  Interventions: Other: perception of vertical after static roll-tilt over 5min

INTERVENTIONS:
Other: perception of vertical after static roll-tilt over 5min — subjects will indicate perceived direction of vertical after 5min of static whole-body roll-tilt.

SUMMARY:
The long-term goal of this research is to advance our knowledge of how the brain combines the information of multiple sensory systems coding for spatial orientation and how adaptation to vestibular imbalance influences spatial orientation. In healthy human subjects verticality perception is accurate while upright. After prolonged roll-tilt, humans show a systematic bias in perceived direction towards the previous roll-tilted position (so-called "post-tilt bias"). Here we evaluate different potential explanations for this bias using both vision-dependent and vision-independent paradigms of verticality perception.

ELIGIBILITY:
Inclusion Criteria:

1. ages 18-65 years
2. informed consent
3. absence of exclusion criteria

Exclusion Criteria:

1. peripheral-vestibular deficit
2. disturbed consciousness
3. history of sensory deficits
4. visual field deficits
5. other neurological or systemic disorder which can cause dementia or cognitive dysfunction
6. intake of antidepressants, sedatives, or neuroleptics
7. pregnancy, unless excluded by a negative pregnancy test
8. known neck pain or status post neck trauma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06-01; Primary Completion 2016-07-01 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Adjustment errors and trial-to-trial variability as assessed by line adjustments (subjective visual vertical (SVV)), adjustments of a rod (subjective haptic vertical (SHV)) or self-adjustments (subjective postural vertical (SPV)) after prolonged roll | measurements will be obtained over periods of 5min in a single session and day
  In all three paradigms (SVV, SHV and SPV) the percept of direction of gravity will be assessed. Parameters will be adjustment errors ("accuracy") and trial-to-trial variability ("precision") based on repetitive adjustments of a luminous line (SVV) or a rod (SHV) after returning to upright position after a period of 5min in static roll-tilt at 90° left-ear down or right-ear down. During the roll-tilt period subjects remain either in the dark or observe a rotating optokinetic (random dot) pattern. Individual mean values and standard deviation (SD) will be calculated for all conditions. Adjustments with the joystick (SPV) will start from 90° ear-down positions after 5min of static roll.

SECONDARY OUTCOMES:
Impact of a rotating optokinetic stimulus (velocity 60°/s) on adjustment errors as assessed by the SVV, the SHV or the SPV after 5min of static roll-tilt at +/- 90° roll. | measurements will be obtained over periods of 5min in a single session and day
  During the 5min period with static roll at +/- 90deg ear-down positions subjects will be presented a rotating optokinetic stimulus (random dot pattern, clockwise or counter-clockwise rotation) in some conditions. Adjustment errors and trial-to-trial variability of conditions with the optokinetic stimulus will be compared to those without the optokinetic stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Straumann, MD, Principal Investigator — University of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No